CLINICAL TRIAL: NCT00028080
Title: Evaluation, Treatment, and Follow-up of Patients With Lyme Disease
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020055; 02-I-0055
Record Dates: First submitted 2001-12-11; First posted 2001-12-12 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-03-31

CONDITIONS: Lyme Disease
Keywords: Borrelia Burgdorferi; Lyme Disease; Infection; Therapy; Natural History; Lyme
MeSH Terms: conditions — Lyme Disease; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lyme Disease: Participants who have been diagnosed with or are strongly suspected to have Lyme disease.

SUMMARY:
This study is designed to establish a population of patients with Lyme disease for evaluation, treatment and follow-up to learn more about the infection.

Patients with active Lyme disease may be eligible for this study.

Participants will have a medical history and physical examination and diagnostic evaluations as appropriate to their individual condition. Laboratory tests may include routing blood and urine tests, X-rays, or other imaging studies, body fluid or tissue cultures, skin biopsy and tests for allergic or immune responses. Treatment will include only medications approved by the Food and Drug Administration, given according to accepted dose schedules and ways of taking the medicines. All diagnostic tests and treatments will be according to standard medical practice for the disease. No experimental procedures will be offered under this protocol.

Patients will be followed as needed for evaluation and treatment of their condition. In general, they will be asked to return at the end of therapy, then 3, 6 and 12 months later, and then every 6 to 12 months. More frequent visits may be required or less frequent visits may be allowed, depending on the individual s condition.

Participants may be asked to undergo the following additional procedures for research purposes:

* Extra blood draws to study Lyme disease and other inflammatory conditions. Blood will be drawn from arm veins. The total amount drawn during any 6-week period will not exceed 450 cc (30 tablespoons) for adults and 7 cc (1/2 tablespoon) per kilogram (2.2 pounds) of body weight for children under 18 years of age.
* Leukapheresis to collect large numbers of white blood cells. Whole blood is collected through a needle in an arm vein, similar to donating blood. The blood circulates through a machine that separates it into its components, and the white cells are removed. The rest of the blood is returned to the body through the same needle. Only adults 18 years of age and older will be asked to undergo leukapheresis.

DETAILED DESCRIPTION:
Lyme disease is a multisystem illness caused by the spirochete Borrelia burgdorferi and it is the most common vector-borne illness in the United States. This protocol is designed to offer evaluation, therapy and follow up to patients with Lyme disease. This is a natural history study, which has the objective of developing a rigorously defined population of patients with Lyme disease to serve as the basis of research in multiple aspects of the infection. These research sub-projects have emphasis in exploring the biological markers of Borrelia infections, assessment of clinical course and outcomes of patients with Lyme infection, and the immunological response to B. burgdorferi infection.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Clinical diagnosis of active Lyme disease at the time of the initial NIH evaluation based on the CDC case definition. Study physician will review history to confirm probable cases.
* Subjects must maintain a private physician for non-protocol related medical complaints and for emergency medical treatment required for these or other of their disorders.

EXCLUSION CRITERIA:

* Post treatment Lyme disease syndrome.
* Unacceptably poor compliance, which, in the opinion of the investigator, would interfere with one's ability to study or provide quality medical care for the patient.

ELIGIBILITY CRITERIA TO UNDERGO APHERESIS:

* Age 18 years or above.
* Weight greater than 110 pounds.
* No known heart, lung, kidney disease, or bleeding disorders.
* Negative HIV, HCV and HBsAg serologies.
* Female subjects should not be pregnant or nursing.
* Patients will have a CBC performed up to 2 weeks before the procedure. In order to be able to undergo the procedure, patient must fulfill all of the below:

  * Hemoglobin greater than 11 g/dL for males and greater than 10 g/dL for females.
  * Platelets greater than 150 k/mm(3).
  * WBC greater than 3.5 x 10(3) uL.
  * MCV above 80.

Women who are able to conceive children must have a negative pregnancy test within 2 weeks before the procedure.

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2002-01-16 (Actual)

PRIMARY OUTCOMES:
Develop a defined population of patients with Lyme disease to serve as the basis of research in multiple aspects of the infection. | 12/31/2030
  Explore the biological markers of Borrelia infections, assessment of clinical course and outcomes of patients with Lyme infection, and the immunological response to B. burgdorferi infection.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana R Marques, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is know yet known if the results of the study will warrant sharing IPD.

REFERENCES:
- [Background] Marques AR. Lyme Neuroborreliosis. Continuum (Minneap Minn). 2015 Dec;21(6 Neuroinfectious Disease):1729-44. doi: 10.1212/CON.0000000000000252. PMID 26633786
- [Background] Wills AB, Spaulding AB, Adjemian J, Prevots DR, Turk SP, Williams C, Marques A. Long-term Follow-up of Patients With Lyme Disease: Longitudinal Analysis of Clinical and Quality-of-life Measures. Clin Infect Dis. 2016 Jun 15;62(12):1546-1551. doi: 10.1093/cid/ciw189. Epub 2016 Mar 29. PMID 27025825
- [Background] Marques AR. Laboratory diagnosis of Lyme disease: advances and challenges. Infect Dis Clin North Am. 2015 Jun;29(2):295-307. doi: 10.1016/j.idc.2015.02.005. PMID 25999225
- [Derived] Gwynne PJ, Clendenen LH, Turk SP, Marques AR, Hu LT. Antiphospholipid autoantibodies in Lyme disease arise after scavenging of host phospholipids by Borrelia burgdorferi. J Clin Invest. 2022 Mar 15;132(6):e152506. doi: 10.1172/JCI152506. PMID 35289310
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2002-I-0055.html